CLINICAL TRIAL: NCT00368888
Title: Clinical Study of New Urine Collection Bag for Infants.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bergaliden Barnavårdscentral (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LIVI4099
Record Dates: First submitted 2006-08-28; First posted 2006-08-29 (Estimated); Last update posted 2006-09-12 (Estimated); Status verified 2006-09

CONDITIONS: Urinary Tract Infection
MeSH Terms: conditions — Urinary Tract Infections

INTERVENTIONS:
Device: Urine collection bag for infants

SUMMARY:
To determine whether a new urine collection bag for infants produces a reliable urine sample for culturing in respect of contamination rate with skin bacteria.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children.

Exclusion Criteria:

* Current infection of any kind. History of urinary tract infection.

Ages: 0 Years to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Dates: Start 2004-03; Study Completion 2006-09

CONTACTS AND LOCATIONS:
Overall Officials: Markus Perlhagen, Doctor, Principal Investigator
Locations (1):
- Bergaliden Barnavårdscentral (Child Care Center), Helsingborg, Sweden